CLINICAL TRIAL: NCT06889025
Title: Electric and Physiological Markers, Underlying Mechanisms and Modulation of Cognitive Functioning and Therapeutic Improvement in Response to tACS/CBTp (Transcranial Alternating Current Stimulation Applied at the Beginning of the Cognitive Behavioral Therapy for Psychosis Session) in Combination With the Usual Pharmacological Treatment in Schizophrenia
Brief Title: Therapeutic Improvement in People With Schizophrenia Undergoing tACS/CBTp (Transcranial Alternating Current Stimulation Applied Pre-cognitive Behavioral Therapy for Psychosis) Associated to Usual Medication Regimen
Acronym: tACS/CBTpSZ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Felicia Iftene (Other)
Collaborators: Providence Care Hospital - Providence Care (Unknown); Queen's University (Other)
Responsible Party: Sponsor-Investigator, Felicia Iftene, Dr. Felica Iftene, Associate Professor, Department of Psychiatry, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB File No: 6044118; TRAQ DSS file - #6036290 (Other Grant/Funding Number: Queen's University)
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; tACS; CBTp
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Mandatory Non-Experimental Procedures:
  16 individual-basis (with duration of 50 minutes), weekly sessions (a form of talk therapy named cognitive behavioral therapy for psychosis) and a booster session of CBTp at each follow up (one month and three after intervention).
  Mandatory Experimental Procedures The tASC with gamma band electric stimulation for 20 minutes at the beginning of the CBTp session is considered experimental and will only be done as part of this study.
  The combination of tASC and CBTp intervention will be applied to the two different groups: one with gamma band electric stimulation for 20 minutes at the beginning of the CBTp session and another group with sham tACS/CBTp (the tACS is sham, but the CBTp is intervention).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tACS/CBTp, both active/ intervention (Experimental): n=14; participants living with schizophrenia/schizoaffective disorder, stable under their usual medication; tACS (gamma band electric stimulation) will be applied the first 20 minutes of the CBTp session (then the device remains in place, but the electric stimulation will be automatically stopped). The CBTp will continue up until a total of 50 minutes/session.
  Interventions: Other: Experimental: tASC/CBTp: gamma band electric stimulation for 20 minutes at the beginning of the CBTp session
- Sham tACS and CBTp (only CBTp active, intervention) (Sham Comparator): n=14, same diagnosis population, gender and age matched; sham tACS, CBTp for 50 minutes/session.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Other: Experimental: tASC/CBTp: gamma band electric stimulation for 20 minutes at the beginning of the CBTp session — For the transcranial stimulation we will use the tES device from NeuroMyst,. The gamma pulses are delivered to a study participant via stimulating electrodes positioned at participant's head according to the required technique. The tACS will be applied the first 20 minutes from the classic CBTp session for the experimental group.
  Arms: tACS/CBTp, both active/ intervention
Other: Sham Comparator — For the Sham group the investigators will use the same tES device from NeuroMyst. The Sham stimulation will be applied only for a few seconds in Sham group. The CBTp will follow the same protocol for both arms.
  Arms: Sham tACS and CBTp (only CBTp active, intervention)

SUMMARY:
The investigators are proposing a new, non-invasive therapeutic model using transcranial alternative current stimulation (tACS), to augment cognitive behavioral therapy for psychosis (CBTp) efficacy in individuals with schizophrenia (SZ). Using EEG brain oscillation activity, as a biomarker of the progression of cognitive deficits in SZ, the investigators aim to understand if addressing the oscillation perturbations could reduce the cognitive deficits. The investigators are using heart rate variability (HRV) as a biomarker of improvement of somatic and mental health. The investigators are aiming also for an analysis through a GBA+ lens, by using along with specific tests for psychosis (PANSS, NSA-16, etc.), the BEM Sex Role Inventory. Considering that cognitive and emotional status is gender dependent, the investigators expect that the therapeutic response could be gender specific. This is a prospective, randomized, repeated-measures, single-blind study design. Pre-intervention, eligible participants will be randomly assigned to one of two treatment arms. Arm 1 (tACS/CBTp n=14); Arm 2 (sham tACS/CBTp, n=14; tACS is sham, but CBTp is active). Intervention (16 weeks): participants in Arms 1 and 2 will receive once weekly tACS/ CBTp or sham tACS/CBTp. Post-intervention: follow-up visits at 4- and 12-weeks post-intervention (with a tACS/CBTp booster session provided each time). The chart review will search for: comorbid metabolic conditions, lab work abnormalities (glycemic level, Hb A, cholesterol), substances use, BMI, type of medication, side effects. Expected outcomes: Participants in Arm 1 will show a better improvement in psychosocial assessment scores, electrical brain activity (tendency to organize the neural oscillations in the gamma frequency range, mainly in frontal lobes) and heart activity (increased HRV). The timeline for recruitment, treatment and follow-up, is 18 months, followed by six months for data analysis, dissemination activities. Population: Individuals with SZ (DSM V criteria) stratified by age and sex. The investigators expect 150 potentially eligible patients from PCH-MHS, with 28 participants consenting to participate.

DETAILED DESCRIPTION:
Rationale. 1% Canadians suffer from Schizophrenia (SZ), a neurodegenerative condition with a high rate of relapse, and important personal, familial and social burden, involving a high cost for care. The suicide rate for people with schizophrenia is over 20 times higher than the general population. While there is no cure, programs and treatments are available to help manage symptoms; however, these have limitations. 60% of patients with SZ do not respond adequately to treatment with medication alone (currently the primary, and often only approach). When CBT for Psychosis (CBTp) is used alongside medication, some improvements have been observed but the debilitating negative symptoms remain (such as reduction of emotional expression, lack of social involvement, inability to initiate goal-directed activities, etc.), which are key factors in long-term disability. A new treatment, transcranial alternating current stimulation (tACS) has therapeutic results in Alzheimer's.

The investigators propose combining these two therapies (CBTp and tACS), in a novel way to increase the overall improvement of negative symptoms in people living with schizophrenia.

Rationale: schizophrenia is characterized by abnormalities in neural circuitries resulting dysfunctional cognition and behavior. Recent randomized double blind clinical trials of tACS in Alzheimer's disease showed a significant improvement in memory performance, along with restoration of intracortical connectivity, as compared to sham tACS. The investigators propose similar cognitive enhancements in people living with schizophrenia. This technique has never been applied before in our studied population and has never used in combination with CBT.

Methodology. Description of intervention: CBTp: 16 individual-basis, 50 minutes length, weekly sessions (CBTp intervention) and 2 booster CBTp sessions at follow up visits (at one month and three months after intervention). tASC/CBTp: two different groups, one with gamma band electric stimulation for 20 minutes at the beginning of the CBTp session (after the first 20 minutes of brain stimulation the tACS device automatically stops and the device remains in place, while the CBTp session continues to run for 30 more minutes) and another group with sham tACS/CBTp (tACS is sham, but CBTp is intervention). For each group the investigators will follow the same protocol.

Number of visit (V): V. 1 (screening, week 0=W. 0); V.2 (enrollment/baseline, W.2, followed by starting intervention); V. 3 (Intervention Session 8/mid-term, W.9); V.4 (End of Intervention W. 17); V.5 (follow-up 1, W.21); V.6 (follow-up 2, W.29). Measures: Primary outcome measures/dependent variables: PANSS, Negative Symptom Assessment, Cognitive Flexibility Scale. Secondary physiological measures: EEG data and HRV: baseline, and end of intervention visit. Secondary psychological measures (WHO Disability Assessment Scale, Brief Betrayal Trauma Survey, BEM Sex Role Inventory Perceived Stress Scale, Working Alliance Inventory, Quality of Life and Enjoyment Scale, STROOP Color and Word test and Personal Evaluation in Transition of Treatment Scale). Eligibility screening measures: EEG; Columbia Suicide Severity Rating Scale; MOCA (over age 65): at screening. The chart review, performed at screening will help with selecting eligible participants. Statistical analysis plan: on SPSS, version 29, main tests will include repeated measures, mixed design analysis of variance and t-tests for two-group comparisons.

Analytical plan. This is a pilot study, and a sample size calculation is usually not necessary (however, there is a basic rule of 12 per group). Our primary focus is estimating average values and variability for planning larger subsequent studies. The investigators will consider all our clients (PCH_MHS) that meet diagnosis criteria (DSM V-TR) and are willing to be included to participate. Estimated sample size: N 150 (age/gender balancing target 75 female and 75 male); after screening the investigators estimate that the final number of participants will be 28, randomly assigned to one of the two intervention groups, following the same protocol (16 weekly tACS/CBTp intervention sessions, plus two booster sessions at the two follow-ups), but the intervention will be different, including sham tACS/CBTp and tACS/CBTp, respectively.

Objectives. Main objective: to elicit cognitive readiness, and therapeutic engagement as well as a better level of functioning and quality of life by adding tACS at the beginning of the CBTp session in participants living with schizophrenia, expecting at the endpoint an improvement in selected psychiatric and psychosocial assessment scores. A sham tACS condition, will ensure quality comparisons for the study group.

The investigators are using EEG brain oscillation activity as a biomarker of the progression of cognitive deficits in schizophrenia, and heart rate variability (HRV) as a biomarker of improvement of somatic and mental health. The investigators are aiming also for a sub-group analysis through a GBA+ lens, by using along with specific tests for psychosis (PANSS, NSA-16, etc.), the BEM Sex Role Inventory.

The investigators don't have healthy controls included in our study populations. Participants in one of the two intervention groups will not receive the current stimulation, but a placebo/sham tACS (the tACS is placebo but the CBTp is the intervention). Not receiving the low electric stimulation that may augment their response to psychotherapy (CBTp), their condition might not improve. The previous studies using only CBTp as intervention reported improvement of the illness (they will receive CBTp anyways). However, these study participants will continue their usual treatments, including antipsychotic treatment.

Devices. For measuring the Heart Rate Variability (HRV), the investigators will use an arm heart monitor. For the transcranial stimulation the investigators will use the tES device from NeuroMyst, featuring tDCS, tACS, tPCS, tRNS and tRCS waveforms as well as blind and double-blind placebo (sham) modes. Using advanced micro-electronics ensures accurate stimulation. Impedance changes can be detected and correct in 50 µ seconds. This means target current levels are super-accurate and super-stable, coming with an adjustable stimulus current of 0 up to 5 mA, with 25 µA increment and adjustable stimulation duration of 15 up to 40 min, with 5 s increment, as well as a study mode for sham stimulation. The electronic unit is intended to generate the electrical pulses of specified waveform, duration and repetition rate. The pulses are delivered to a study participant via stimulating electrodes positioned at participant's head according to the required technique. tES is an Investigational Device Exemption, with low risk for participants, that adhere to the international safety and recommended FDA guidelines.

Questionnaires. Study staff will ask each participant to answer questions in order to complete the study specific scales and assessments to check cognitive (mental) function, how well they are able to perform daily activities, their motivation and symptoms of schizophrenia status. Some of the questionnaires/assessments are self- assessments completed on paper; others will be completed by an interviewer (research staff). Trained study staff will give instructions on how to complete all of the questionnaires/ assessments. The participants will be allowed to take short breaks during these assessments if they need them. For some of the questionnaires/assessments, the participants should hold certain medications such as sleep or allergy medications (in particular benzodiazepines used to treat anxiety) at least 8 hours before the study visits. The study staff will tell them (before these visits) which medications should not be taken, if this applies to them. Some of the questionnaires/assessments must be done at approximately the same time of day. This is very important, and if the study participants are not able to arrive at the clinic on time for these visits, then the study staff may need to re-schedule the visit with them for another day. During the study visits the participants will be asked about their life experiences (positive and negative), relationships, and mental state (emotions, thoughts, feelings, symptoms); about their current experiences and problems they may be having, and information about their personal experience of schizophrenia, as this relates to the illness, stigma, its effects on their daily life such as stressors; about how they perceive their illness, about things that improve and worsen how they feel, and about their activities/events that they participate in or perceive around them. The names of the scales used in this study are: PANSS, Negative Symptom Assessment (NSA), Cognitive Flexibility Scale (CFS), WHO Disability Assessment Scale (WHODAS), Brief Betrayal Trauma Survey (BBTS), Perceived Stress Scale (PSS), Working Alliance Inventory (WAI), Quality of Life and Enjoyment Scale (QOL), STROOP Color and Word test, Columbia Suicide Severity Rating Scale (C-SSRS), BEM Sex Role Inventory and Personal Evaluation in Transition of Treatment Scale (PETIT), Montreal Cognition Assessment (MoCA) (over age 65).

The chart review at screening will help with selecting eligible participants. The chart review will search for: comorbid metabolic conditions, lab work abnormalities (glycemic level, Hb A, cholesterol), substances use, BMI, type of medication, side effects. Any chart reviews will be conducted by hospital-appointed individuals who have the privilege to access this information.

Sample size. This is a pilot study, and a sample size calculation is usually not necessary (however, there is basic rule of 12 per group). The investigators will consider all our clients (PCH-MHS) that meet diagnosis criteria (DSM V-TR) and are willing to participate. Our primary focus is estimating average values and variability for planning larger subsequent studies. Estimated sample size: N 150 (age/gender balancing target 75 female and 75 male); after screening the investigators estimate that the final number of participants will be 28, randomly assigned to one of the two intervention groups. The intervention groups will follow the same protocol (16 weekly intervention sessions with two follow-ups), but the intervention will be different, including sham tACS/CBTp and tACS/CBTp, respectively.

Recruitment. A letter and a poster will be distributed to psychiatrists at Providence Care Mental Health Services (PCH-MHS), informing them they can refer clients to the CBTp Clinic and they are invited to refer potential participants that meet an inclusion/exclusion criteria. Word of mouth and brochures/flyers will be prepared. The clinic staff or directly the participant will then contact our Research Coordinator/Assistant to communicate more information to the potential participant.

All participants included will have a diagnosed mental health disorder of schizophrenia or schizoaffective disorder. The investigators plan to include individuals who are both inpatients and outpatients at Providence Care Hospital. This includes participants who may be in long-term care. Potential participants in the study will be referred to the CBTp Clinic at Providence Care Hospital by the participant's primary treating psychiatrist. The treating psychiatrist will explain verbally and in writing that the referral is completely optional and that participation in any related study is entirely secondary and completely optional. During the first meeting at the CBTp Clinic, the potential participant will be informed about the study. The potential participant will be informed that their participation in the study is entirely optional alongside the standard clinic disclosures about privacy/confidentiality. They will have an opportunity to consider further involvement in a study by being given a break if they decide between meeting clinic personnel and being proposed written consent. Express written consent to participate in the study will be obtained by a member of the research team who is not in the circle of care of the participant (at arm's length). Participant withdrawal forms have been created to document any withdrawal accurately.

DISABILITY: Individuals will be excluded if they have severe or moderate intellectual disability or dual diagnosis, due to the nature of CBTp, that requires the learning of coping strategies, adequate attention and memory, engagement using speech, and appreciation of consequences of action, thoughts, behaviors, emotions, and beliefs which are limited in severe intellectual disability.

LANGUAGE AND LINGUISTIC PROFICIENCY: Individuals will be excluded if they do not have ability to understand English with reading level at or above grade 6. The ability for an individual to meaningfully engage in a CBTp talk therapy would be limited if their English level is limited to a grade 6 level and is thought to not be substantially beneficial to the individual.

AGE: Participants recruited will be included if they are aged 18-65. Individuals older than 65 years of age will be required to be assessed by the Montreal Cognitive Assessment and will be included in the study if results validate adequate cognitive performance. The Montreal Cognitive Assessment will be administered at the screening stage (score under 26 will be exclusion criteria).

Inclusion criteria. Individuals, with at least 5 years duration of illness, that meet diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual for Mental Disorders-5 and at least one residual positive symptom (as determined by the referring physician); no change in medication regimen for at least 1 months (minor dose adjustments and/or change in medication involving symptoms as sleep, anxiety or medical symptoms such as fever, pain, are permitted); persons of all genders between ages 18-65 (participants 65+ may be eligible depending on performance on cognitive assessment); ability to understand English with reading level at or above grade 6; able to understand and comply with the requirements of the study; provision of written informed consent.

Exclusion criteria: current illicit drug substance abuse; current suicidal ideation; current enrollment in CBTp or other formalized psychosocial interventions; undergone vagotomy or surgery upon the vagus nerve; comorbid neurological condition; severe or moderate intellectual disability; currently undergoing hormone therapy; under age 18; changes in medication/new hospitalization for worsening symptoms and/or presence of suicidal ideation. NOTE: for the last exclusions, these are no longer exclusion criteria for subjects that have passed visit 5, end of intervention, during follow-ups stage; however, the results of the follow-up visits will count at the final results, depending on the severity/imminent danger of symptoms and medication changes, at the best judgment of the principal investigator.

Patient care considerations. The main standard of care is medication management for adults with schizophrenia/schizoaffective disorder. When an individual requires other services or care, generally a referral is made to obtain these services. A proportion of adults with schizophrenia in the community may also have social or skill support via a community treatment team. The research Lab is situated in a hospital setting which is well resourced to support care in case of an emergency on site. Participants will be receiving their standard usual care throughout the study.

Premature withdrawal or suspension may occur if imminent safety concerns are disclosed to a study team member or a member of the CBTp Clinic by the participant. Withdrawal would be considered with the best interests and safety of the participant considered and foremost. An example of this would be if a participant indicated suicidal or homicidal ideation with a plan to carry out such an act at any point in time. After safety considerations are met and satisfied, the participant would be eligible to return or be included in the study.

The research team may temporarily or fully stop the study if there is any reason to believe that there is a medical reason why a participant may need to stop the study. Some of the reasons why this might happen are listed below: • their condition worsens or does not improve, and their doctor thinks they need a different treatment. • the study treatment or procedures are found to be unsafe or ineffective. • they are unable to follow instructions given to them about the study, or they otherwise cannot do or continue to do what they need to in order to participate in the study. • they develop another serious disease. • they become pregnant. • cancellation by the sponsor or regulatory authority, or for other unforeseen reasons that make it necessary to stop their study participation. If a participant is removed from the study from the study, the study doctor will explain to them why the participant was removed. A participant may also be temporarily suspended or stop their participation in the study in the event they require attention if it is believed there is a risk of harm to themselves or others. This may be indicated by a member in their circle of care or them or by the clinician-researchers on the team. In the event there is a risk of harm to themself or others, after the risk is no longer deemed significant, they may be able to continue the study.

Inform consent procedure. Potential participants will first verbally consent for their contact information to be shared with a Research Coordinator/Assistant to be contacted about the study, and to learn more about the study prior to agreeing to participate. A Research Coordinator/Assistant will contact the potential participant and arrange a meeting to discuss the study. At the meeting with the Research Coordinator/Assistant, the potential participant will learn about the study and will verbally be informed about content on the ICF form. The Letter with ICF will be presented and explained portion by portion, with the Research Coordinator/Assistant. The Research Coordinator/Assistant will allow the participant time, if they opt, on their own to review the form for 10 minutes, if they desire. They can even take home an unsigned document to ask for advice from their family, family physician, etc. If the participant agrees to proceed, they will be asked for their express written consent. Written consent will be re-assessed directly prior to undertaking the task. After this time, an appointment will be arranged for a screening visit. At each stage throughout the participants' engagement in the study, researchers will ask for verbal consent to continue. At this time, a participant will be told they have a choice to proceed or assess their willingness to participate. It is also foreseeable that if a participant comes to their respective appointments with the research team at subsequent points, willingness to participate will be implied. If a participant elects to withdraw from any aspect of the study, then, the research team has created a system to note participant withdrawal and how this was obtained for record-keeping reasons.

There are members of the research team who will be considered within the direct circle of care of the potential participant; where this is so, a member of the research team outside the direct circle of care of the potential participant will be designated as the individual to obtain written consent and also the individual who the participant can contact if the potential participant would like to withdraw/discontinue further participation. This arrangement will uphold the voluntary nature of consenting and minimize undue influence or power imbalance.

Where a participant has difficulty reading, a member of the research team will verbally communicate the information on a form/questionnaire if a participant requires clarification. Every effort will be made to try to help eligible participants with communication difficulties.

In this study the investigators don't enroll participants incapable to sign informed consent. To proactively monitor changes in the status of capacity, mid-way through the study, the research team will seek confirmation of the capacity status of the participant from healthcare personnel. As is typical ethical practice outside the scope of this study, if members of the CBTp Clinic (by way of observation/professional judgment) suspect a change in capacity in the participant, the participant's primary treating psychiatrist will be notified, and a re-assessment would take place.

Reimbursement. The investigators will give each participant $10 reimbursement to cover out-of-pocket expenses such as meals and parking for each of the 6 visits that are required as part of the study. Payments will be provided after each task is complete.

Some participants may incur expenses for food and travel (bus). Participants will be encouraged to bring a lunch or snack with them, as indicated on the ICF in light of this. The compensation will cover costs of bus transportation.

Potential risks. Transcranial alternative current stimulation: There are risks to taking part in any clinical study. If they receive a placebo/sham tACS, they will not receive the electric stimulation that may augment the response to psychotherapy (CBTp). If they receive active tACS before psychotherapy, then side effects may occur. Some of the side effects that may occur during this study can be treated. The adverse events are: very mild tingling sensation, fatigue and a light itching skin sensation under the stimulus, mild headache, dizziness, all these disappearing just after stimulation. With tACS no persistent adverse events have been reported, but the adverse events of the repetitive tACS application have not been fully clarified. In this type of stimulation technique, no serious adverse effects were reported.

Questionnaires: Some questionnaires may ask about stressful events in their life which may cause to them feel discomfort or remember things that may have upset them in their past. If they feel the content of a questionnaire is distressing, they are encouraged to let the study coordinator know at the time or at any later time. A member of research team can discuss this with them and refer this to a member of their care team whom they identify and consent to (the investigators will ask them for written consent to disclose this information if they decide). The participant's name will never be placed on a questionnaire to maintain their own privacy and to protect their confidentiality, and if they write their name by accident, a sticker that cannot be removed easily containing their participant ID will be placed over this to maintain their privacy. The participants may also feel frustrated or confused by language in the questionnaires. If there are words in any written material or things the investigators explain that require more clarify for them, members of the research team will be pleased to help them and clarify details to their satisfaction.

Data security and scientific advancements: Even with data security protections in place, there is a risk that participant information could be released by accident.

The plan to mitigate the risk of psychological or emotional risk will be managed by the research team, and training interviewers to administer questionnaires to be thoughtful, sensitive, and cognizant of the types of questions they are asking and anticipating these effects and potential thought processes the participants may experience. These are essential strategies to ensure sensitive and polite communication and help researchers learn how to read verbal and non-verbal communication that may communicate discomfort. In case of a confidentiality breach, in spite of the safeguards in place, the investigators will immediately take steps to contain it, notify the participant, investigate and remediate.

The chart review will search for risk factors that may influence the participant response to study intervention: comorbid metabolic conditions, lab work abnormalities (glycemic level, Hb A, cholesterol), substances use, BMI, type of medication, side effects. Only personnel with designated hospital appointments (Departmental Assistant Status/Departmental Research Assistant Status at Providence Care Hospital) or physicians at Providence Care Hospital who are part of the research team will have access to any Personal Health Information. The access will be necessary to corroborate information given during Interviewer-Administered Interviews linked with questionnaires.

Access to medical records and/or study data will be limited to authorized personnel. Electronic data will be stored on a hospital or other institutional network with firewalls and other security and back-up measures in place. Data stored on laptops or mobile devices will be encrypted. Paper copies of study data will be stored in locked filing cabinets in a secure location.

Dr. Felicia Iftene, A. Farcas will have access to data. Data will be stored 15 years under participant ID numbers (anonymized) on the electronic data will be stored on a hospital or other institutional network with firewalls and other security and back-up measures in place.

Any data that exists in identifiable form (Name) will immediately, at first opportunity, be converted and replaced with participant ID. A Master-List of code-linking identifiers will only be held by Dr. Iftene, A. Farcas for 15 years after the end of study.

Data collected on paper, with the exception of the consent form, will be anonymized. Data collected on paper will be stored in the archive, in locked filing cabinets at Providence Care Hospital. The data will be kept for 15 years in a de-identified format, in the archive.

Impact Novelty and innovation. Our goal is to find solutions to improving treatment trajectories for individuals suffering from schizophrenia. With this study, the investigators will be the first to examine the possibility of augmenting the efficacy of CBTp by inducing neural oscillations within the gamma range add-on to the CBTp session, contributing new knowledge to literature.

Clinical benefit. 28 clients will have the opportunity to benefit from our CBTp intervention with or without tACS.

Social costs. The new type of intervention will allow for personalized and highly impactful treatment. This will lead to quality-of-life improvement for participants as well as for support members (family and caregivers) and will reduce health care costs.

Dissemination. The investigators anticipate publishing up to 5 new peer reviewed publications and present the results to different scientific events. This pilot study will generate a data set that will support future grant application.

Education. Two master students from the Center for Neuroscience Studies, are working on this project, under the supervision of Dr. Iftene and Dr. O'Brien.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals, with at least 5 years duration of illness, that meet diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual for Mental Disorders-5 and at least one residual positive symptom (as determined by the referring physician);
2. no change in medication regimen for at least 1 months (minor dose adjustments and/or change in medication involving symptoms as sleep, anxiety or medical symptoms such as fever, pain, are permitted);
3. all genders between ages 18-65 (participants 65+ may be eligible depending on performance on cognitive assessment);
4. ability to understand English with reading level at or above grade 6;
5. able to understand and comply with the requirements of the study;
6. provision of written informed consent.

Exclusion Criteria:

1. current illicit drug substance abuse;
2. current suicidal ideation;
3. current enrollment in CBTp or other formalized psychosocial interventions;
4. undergone vagotomy or surgery upon the vagus nerve;
5. comorbid neurological condition;
6. severe or moderate intellectual disability;
7. currently undergoing hormone therapy;
8. under age 18.

NOTE: changes in medication/new hospitalization for worsening symptoms and/or presence of suicidal ideation are no more exclusion criteria for subjects that have passed visit 5 (end of intervention, during follow-ups stage); however the results of the follow-up visits will count at the final results, depending on the severity/imminent danger of symptoms and medication changes, at the best judgment of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
PANSS (Positive and Negative Symptoms of Schizophrenia Scale) | Positive and Negative Symptoms of Schizophrenia scale will be applied at: Visit 1, Screening (Week 0); Visit 4, End of intervention (Week 17); Visit 5,Follow-up 1 (Week 21); Visit 6 Follow-up 2 (Week 29).
  The PANSS is a standardized clinical interview that rates the presence and severity of positive and negative symptoms and general psychopathology for people with schizophrenia within the past week. The scale consists of 30 items: seven positive, seven negative, and 16 general psychopathology symptoms. The symptom severity for each item is rated according to a 7-point scale (1 = absent; 7 = extreme) to best describe the symptom's presentation. The clinical interview takes approximately 45 minutes. The patient is rated from 1 to 7 on 30 different symptoms based on the discussion and reports of family members or primary care hospital workers. As 1 is the lowest score for each item, a patient can not score lower than 30 for the total PANSS score. Scores are often given separately for positive items, negative items, and general psychopathology.
NSA-16 (Negative Symptom Assessment) | Negative Symptom Assessment-16: Visit 2, Baseline (Week 1); Visit 4, End of intervention (Week 17); Visit 5, Follow-up 1 (Week 21); Visit 6 Follow-up 2 (Week 29).
  The NSA-16 assesses the presence, severity, and range of negative symptoms associated with schizophrenia. For rapid clinical assessment or screening of patients for negative symptoms, the NSA-4 was developed as a simplified version, retaining only 4 of the 16 items: restricted speech quantity, reduced emotion, reduced social drive, and reduced interests. Each of the four items and the overall global negative symptoms is rated on a 1 to 6-point scale where '1' represents no reduction from normal behaviors associated with the item and '6' represents a severe reduction in or absence of the behavior, with markedly impaired functionality. With respect to overall accuracy and predictive validity, the NSA-4 is comparable to the NSA-16.
CFS (Cognitive Flexibility Scale) | Cognitive Flexibility Scale: Visit 2, Baseline (Week1 ); Visit 3 Mid point of intervention (Week 9); Visit 4, End of intervention (Week 17); Visit 5, Follow-up 1 (Week 21); Visit 6, Follow-up 2 (Week 29).
  The CFS assesses cognitive flexibility as a factor that facilitates the individual's adaptability towards events. Cognitive flexibility refers to a person's awareness that different communication styles exist in every situation and the person's willingness and self-efficacy to use different communicative styles. The scale has 12 items pertaining to the three elements of cognitive flexibility: a person's awareness of alternative communicative styles, willingness to be communicatively flexible, and self-efficacy in being communicatively flexible. The scale utilizes a 6-point Likert-type scale for each item (with 6 as "strongly agree," 5 as "agree," 4 as "slightly agree," 3 as "slightly disagree," 2 as "disagree," and 1 as "strongly disagree"). The total score was used to calculate a global score ranging from 12 to 72, with questions 2, 9, 11, and 12 being reverse-coded. A higher score indicates higher cognitive flexibility.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | The Heart Rate Variability will be determined at Visit 2, Week 1, before and immediately after the first intervention (tACS/CBTp); it will be determined also pre and post the 16th intervention, Visit 4, Week 17.
  Heart Rate Variability (HRV) refers to the variation in time between consecutive heartbeats, a normal physiological phenomenon indicating the body's ability to adapt to stress and demands. There is no single "ideal" HRV, a higher HRV generally indicates better cardiovascular health and fitness, with a normal range other considered to be between 40 and 100 milliseconds.
  However, individual HRV levels vary based o age, fitness level, and other factors and tracking baseline HRV and trends for an individual, is more important than comparing to others.
Electroencephalogram (EEG) | Electroencephalogram will be performed at the Visit 1, Screening (Week 0) and Visit 5 End of intervention (Week 17) - before and at the end of intervention (the 16 tAC/CBTp sessions)
  Electroencephalogram detects abnormalities in brain waves, or in the electrical activity of the brain. The electrical charges resulting from the activity of the the brain cells, are collected by scalp electrodes, amplified and recorded as a graph on a computer, or printed out on a paper. Our previous EEG recordings showed reduced power and synchronization on gamma oscillations, that in healthy people are 30-100HZ, but in people with schizophrenia gamma activity is narrowly defined as 37-41 Hz. Gamma oscillations specifically controls the connectivity between different specific brain regions, which is crucial for perception, movement, memory and emotions. We are performing resting state EEG (no stimulation, no tasks) an we will analyze the EEG brain oscillation activity, targeting the possible changes of the gamma band activity in the prefrontal cortex (we are looking at the tendency to organize the neural oscillations in the gamma frequency range, mainly in frontal lobes).
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | The WHODAS 2.0 will be performed at: Visit 2, Baseline (Week 1), Visit 4, End of intervention (Week 17), Visit 5, Follow-up 1 (Week 21), Visit 6, Follow-up 2 (Week 29).
  The WHODAS 2.0 measures the level of functioning in six domains of life: cognition - understanding and communicating; mobility - moving and getting around; self-care - attending to one's hygiene, dressing, eating and staying alone; getting along - interacting with other people; life activities - domestic responsibilities, leisure, work and school; participation - joining in community activities, participating in society.
  The 36-item version of WHODAS 2.0 is the most detailed (questions about the difficulties experienced in the past 30 days). It allows users to generate scores for the six functioning domains and calculate an overall functioning score. The average interview time for the interviewer-administered 36-item version is 20 minutes. The simple sum of the scores of the items across all domains constitutes a statistic that describes the degree of functional limitations. The scores are ranging from o to 100, where higher scores indicate greater disability
The Quality-of-Life Enjoyment and Satisfaction Questionnaire Short Form (Q-Les-Q-SF) | The Q-Les-Q-SF will be performed at: Visit 2, Baseline (Week 1); Visit 3 Mid-way intervention (Week 9), Visit 4 End of intervention (Week 17); Visit 5 Follow-up 1 (Week 21); Visit 6 Follow-up 2 (Week 2.9)
  The Q-Les-Q-SF is a 16-item, participant-scored survey utilized to quantify changes in quality of life. The Q-LES-Q-SF evaluates general activities that are assessed in the longer form: physical health, feelings, work, household duties, school/course work, leisure time activities, and social relations. Participants rate their satisfaction using a 5-point scale ranging from 1 (very poor) to 5 (very good). A total score is derived from 14 items, with a maximum score of 70, higher scores indicating greater life satisfaction and enjoyment.
Brief Betrayal Trauma Survey (BBTS) | Brief Betrayal Trauma Survey will be performed at Visit 2, Baseline.
  The Brief Betrayal Trauma Survey - BBTS is a semi structured interview, that measures 14 potentially traumatic events involving mistreatment by someone close, not so close, and non-interpersonal events. Respondents indicate how frequently they experienced an event before and after age 18. Scoring: categorizing of items into High, Medium and Low Betrayal.
Perceived Stress Scale (PCP) | Perceived Stress Scale (PCP) will be performed at: Visit 2, Baseline (Week 1), Visit 4, End of intervention (Week 17), Visit 5, Follow-up 1 (Week 21), Visit 6, Follow-up 2 (Week 29).
  The Perceived Stress Scale (PCP) is one of the most widely used psychological instruments for measuring stress perception. It measures the degree to which situations in one's life are perceived as stressful. The 10 items inquire on how unpredictable, uncontrollable, and overloaded respondents find their lives as well as current levels of experienced stress. The questions in the PSS ask about feelings and thoughts concerning experiences during the last month. In each item, respondents are asked how often they felt a certain way. Individual scores on the PSS can range from 0 to 40, with higher scores indicating higher perceived stress.
The Personal Evaluation of Transitions in Treatment (PETiT). | The Personal Evaluation of Transitions in Treatment (PETiT) will be performed at: Visit 2, Baseline (Week 1), Visit 4, End of intervention (Week 17), Visit 5, Follow-up 1 (Week 21), Visit 6, Follow-up 2 (Week 29).
  The PETiT is a self-administered scale, user-friendly and sensitive to changes associated with treatment over time. Consisting of 30 items, it considers the respondent's health in the last week and offers one of three responses ('often,' 'sometimes,' or 'never'). The scale assesses two highly relevant domains for schizophrenia: adherence-related attitude (includes six items reflecting adherence and feelings towards medication) and psychosocial functioning (24 items describing patient characteristics such as clarity, energy, concentration, functioning, sex drive and memory). The PETiT total score ranges from 0 to 60, with higher scores indicating better patient health-related quality of life.
The Working Alliance Inventory - Short Revised (WAI-SR) - both forms: for client and therapist. | The Working Alliance will be tested at Visit 3, Mid-term through intervention (Week 9) and Visit 4, End of intervention (Week 17).
  The WAI-SR measures three critical aspects of the therapeutic alliance: agreement on the tasks of therapy, agreement on the goals of therapy and development of an affective bond. The 12 items are rated on a 5-point Likert scale ranging from 1 = 'never' to 5 = 'always.' The scores range from 5 to 20, with higher scores indicating a better therapeutic alliance. Completing the WAI-SR takes about 5 minutes.
The BEM Sex Role Inventory (BSRI) | The BEM Sex Role Inventory (BSRI) is performed at Visit 1, Screening (Week 0)
  The BEM Sex Role Inventory (BSRI) is a psychological tool used to measure an individual's perception of their own masculinity and feminity, and it is used to research gender roles, with the understanding that individuals can express both masculine and feminine traits. The interview has 12 items, with scores on a 1 (never or almost never true) -7 (always or always true) scale with average calculated for masculine and feminine traits, and then categorizes them as masculine, feminine, androgynous, or undifferentiated based on those scores. Each item is assigned a category as follows: M for masculine, F for Feminine, N for Neutral.
The STROOP Color and Word Test | The STROOP Color and Word Test will be applied at Visit 2, Baseline (Week 0) and at Visit 4, End of intervention (Week 17).
  The STROOP Color and Word Test, developed by John Ridley Stroop, is a neuropsychological test that measures cognitive interference by asking participants to name the ink color of words, which are printed in a color that conflicts with the word itself.
  The STROOP scores are based on 3 factors: color-naming, interference, and speed, converted into T score for interpretation. A T-score of 40 or less in considered low, while above 40 is considered normal.

OTHER OUTCOMES:
Eligibility Screening Measures: Columbia Suicide Severity Rating Scale | At Screening, Visit 1(Week 0).
  The Columbia Suicide Severity Rating Scale - C-SSRS is a questionnaire developed by multiple institutions, including Columbia University, to help establish a person's immediate risk of suicide. Its questions are phrased for use in an interview format but can be completed as a self-report measure if necessary. The C-SSRS measures four constructs: the severity of ideation, the intensity of ideation, behavior and lethality. It includes "stem questions," which, if endorsed, prompt additional follow-up questions to obtain more information. The C-SSRS comprises ten categories, all of which maintain binary responses (yes/no) to indicate the presence or absence of the behavior. The outcome of the C-SSRS is a numerical score with no specified clinical cut-offs due to the binary nature of the responses to items. Ultimately, interpretation is derived from a thorough clinical assessment, client history, and clinical expertise.
Eligibility Screening Measures: The Montreal Cognition Assessment (MoCA), for participants over age of 65. | The Montreal Cognition Assessment MoCA will be performed at Visit 1, Screening (Week 0), to participants over age of 65 (to exclude a possible cognitive decline).
  The The Montreal Cognition Assessment MoCA is a popular tool used in clinical practice when assessing for mild cognitive dysfunction. This instrument evaluates various cognitive domains, including attention, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. Administering the MoCA takes around 10 minutes, and the total possible score is 30 points. A score of 26 or higher is considered normal, while a final score below 26 suggests mild cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Iftene, Associate Professor, Md, PhD, Principal Investigator — Department of Psychiatry, Queen's University
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is only a small pilot study. If our results will be encouraging we will apply for a larger sample size grant and we will make data available at that point.

REFERENCES:
- [Background] Tsuchimoto R, Kanba S, Hirano S, Oribe N, Ueno T, Hirano Y, Nakamura I, Oda Y, Miura T, Onitsuka T. Reduced high and low frequency gamma synchronization in patients with chronic schizophrenia. Schizophr Res. 2011 Dec;133(1-3):99-105. doi: 10.1016/j.schres.2011.07.020. Epub 2011 Aug 16. PMID 21849245
- [Background] Benussi A, Cantoni V, Cotelli MS, Cotelli M, Brattini C, Datta A, Thomas C, Santarnecchi E, Pascual-Leone A, Borroni B. Exposure to gamma tACS in Alzheimer's disease: A randomized, double-blind, sham-controlled, crossover, pilot study. Brain Stimul. 2021 May-Jun;14(3):531-540. doi: 10.1016/j.brs.2021.03.007. Epub 2021 Mar 21. PMID 33762220
- [Background] Turner DT, Burger S, Smit F, Valmaggia LR, van der Gaag M. What Constitutes Sufficient Evidence for Case Formulation-Driven CBT for Psychosis? Cumulative Meta-analysis of the Effect on Hallucinations and Delusions. Schizophr Bull. 2020 Sep 21;46(5):1072-1085. doi: 10.1093/schbul/sbaa045. PMID 32221536
- [Background] Jones M, McDermott B, Oliveira BL, O'Brien A, Coogan D, Lang M, Moriarty N, Dowd E, Quinlan L, Mc Ginley B, Dunne E, Newell D, Porter E, Elahi MA, O' Halloran M, Shahzad A. Gamma Band Light Stimulation in Human Case Studies: Groundwork for Potential Alzheimer's Disease Treatment. J Alzheimers Dis. 2019;70(1):171-185. doi: 10.3233/JAD-190299. PMID 31156180
- [Background] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819
- [Background] Farcas A, Iftene F. Findings, limitations and new directions in tACS studies in schizophrenia research: A scoping review. J Psychiatr Res. 2022 Jul;151:291-298. doi: 10.1016/j.jpsychires.2022.04.036. Epub 2022 Apr 29. PMID 35525231
- [Derived] Iftene F, Farcas A, O'Brien S, Bowie CR, Best M, Ayonrinde O, Landry T, Carlson J, Davidson S, Rodgerson E, Theis A. Therapeutic Improvement in People with Schizophrenia Undergoing tACS/CBTp (Transcranial Alternating Current Stimulation /Cognitive Behavioural Therapy for Psychosis) Associated with Usual Medication Regimen: Protocol for a Pilot, Randomized, Single-Blind Trial. JMIR Res Protoc. 2025 Nov 21. doi: 10.2196/80593. Online ahead of print. PMID 41273718